CLINICAL TRIAL: NCT03044067
Title: The Effects of Pain Neuroscience Education Plus Exercise in the Management of Fibromyalgia: A Randomized Controlled Trial
Brief Title: Effects of Pain Neuroscience Education in Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Alejandro Luque-Suarez, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniversityMalaga
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-02

CONDITIONS: Fibromyalgia
Keywords: Chronic pain; Fibromyalgia; Pain neuroscience education; Exercise
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain neuroscience education + Exercise (Experimental): Pain neuroscience education can be defined as an educational session or sessions describing the neurobiology and neurophysiology of pain, and pain processing by the nervous system. It will be applied three times (at baseline, one week and one month after intervention). Exercise will be based on a set of 4 exercise implicating flexion, extension, lateral rotation and abduction of lower and upper extremities.
  Interventions: Other: Pain neuroscience education + Exercise
- Exercise (Active Comparator): Exercise will be based on a set of 4 exercise implicating flexion, extension, lateral rotation and abduction of lower and upper extremities. Participants will attend three appointments per week over three weeks. They will complete three sets of 10 repetitions, with the exercises progressed in difficulty at each appointment.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Pain neuroscience education + Exercise — A session of Pain neuroscience education + Exercise covers the activity, strength and endurance of lower and upper muscles of the extremities. Besides that it will be covered the understanding and acknowledgement about how pain is processed.
  Arms: Pain neuroscience education + Exercise
Other: Exercise — A session of exercise covers the activity, strength and endurance of lower and upper muscles of the extremities.
  Arms: Exercise

SUMMARY:
Fibromyalgia is one of the main causes of chronic musculoskeletal widespread pain. This condition presents a global prevalence of 2.7%, and it is more prevalent in women (with a female to male ratio of 3:1) over 50 years of age with low education level and low socioeconomic status, living in rural areas. High direct medical costs and significant indirect costs of this condition can't be ignored.

DETAILED DESCRIPTION:
Study design and setting: The design of the present study will be a randomized controlled trial with 2 follow-ups (one week and one month after intervention) that will be performed between May 2017 and June 2017 in one private clinic in Malaga, Spain. The outcomes will be assessed at baseline (t1), one week after intervention (t2), and one moth after intervention (t3). Written informed consent will be acquired for all participants prior to their participation. The study will be implemented and reported in line with the CONSORT statement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years.
* Willing and able to participate
* Diagnosis of Fibromyalgia

Exclusion Criteria:

* Systemic diseases
* Pain and function due to other rheumatic disorders such as: osteoarthritis, rheumatoid arthritis, ankylosing spondylitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline function at 1 month | 1 month
  This outcome will be measured with the pain disability index (PDI)
Change from Baseline pain at 1 month | 1 month
  This outcome will be measured with the numerical pain rating scale (NRS)

SECONDARY OUTCOMES:
Change from Baseline self-efficacy at 1 moths | 1 month
  Pain Self-Efficacy Questionnaire (PSEQ) contains 10 questions that will be measure the patient's confidence in performing certain activities despite pain.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Luque Suarez, PhD, Principal Investigator — University of Malaga

IPD SHARING:
Plan to Share IPD: No